CLINICAL TRIAL: NCT04912921
Title: Effect of Palmitoylethanolamide on Proinflammatory Markers in Adults Recently Diagnosed With COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STUDY00012462
Record Dates: First submitted 2020-10-15; First posted 2021-06-03 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Inflammation; COVID19
Keywords: palmitoylethanolamide; curcumin
MeSH Terms: conditions — Inflammation; COVID-19 | interventions — palmidrol; microcrystalline cellulose; Curcumin

STUDY DESIGN:
Intervention Model Description: double-blind, randomized, controlled trial
Who Masked: Participant, Investigator
Masking Description: Palmitoylethanolamide and placebo tablets are identical in appearance and presented to participant in unlabeled opaque containers by investigators blinded to container content. Curcumin and control tablets are identical in appearance and presented to participant in unlabeled opaque containers by investigators blinded to container content
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- palmitoylethanolamide (Experimental): Levagen
  Interventions: Dietary Supplement: palmitoylethanolamide
- Placebo (Placebo Comparator): microcrystalline cellulose
  Interventions: Dietary Supplement: Placebo
- HydroCurc (Experimental): curcumin
  Interventions: Dietary Supplement: Curcumin
- Control (Placebo Comparator): microcrystalline cellulose
  Interventions: Dietary Supplement: Control (microcrystalline cellulose)

INTERVENTIONS:
Dietary Supplement: palmitoylethanolamide — 4 tablets taken daily (2 in the am and 2 in the pm)
  Other Names: Levagen
  Arms: palmitoylethanolamide
Dietary Supplement: Placebo — 4 tablets taken daily (2 in am and 2 in pm)
  Other Names: microcrystalline cellulose
  Arms: Placebo
Dietary Supplement: Curcumin — 500 mg HydroCurc® twice a day
  Other Names: Hydrocurc
  Arms: HydroCurc
Dietary Supplement: Control (microcrystalline cellulose) — 2 tablets taken daily
  Other Names: microcrystalline cellulose
  Arms: Control

SUMMARY:
Two randomized controlled trials will be conducted to examine the effect of a food supplement on proinflammatory cytokines and biomarkers in an adult population recently diagnosed with COVID-19 who are asymptomatic or experiencing only mild symptoms. The supplement, palmitoylethanolamide (PEA), is marketed under the trademarked product with increased bioavailability and format versatility: Levagen+™ (Gencor Pacific Limited, Irvine, CA). The supplement curcumin is marketed under the trademarked product with increased bioavailability: HydroCurc (Gencor Pacific Limited, Irvine, CA)

DETAILED DESCRIPTION:
Inflammation is at the core of many chronic conditions and exacerbates infectious conditions, and inflammatory responses appear to be key determinants of the severity of COVID-19 infection. Hence, controlling inflammation is considered a key strategy for slowing the progression of disease and tissue pathology. This research offers a natural, dietary approach to managing inflammation by reducing the mediators of inflammation. The beneficial effects of palmitoylethanolamide (PEA) and for curcumin for reducing inflammation is documented in the research literature. The proposed research will expand this literature in a novel manner. The investigators propose to demonstrate the efficacy of these dietary supplements in individuals from a campus population with robust immune protection - those who recently tested positive for COVID-19 but were asymptomatic or mildly symptomatic. Since a college population is under many stressors which raise inflammatory profiles during the academic year, and since a college population is exposed to infectious agents on campus, maintaining strong protective immune system following a COVID-19 infection is important.

ELIGIBILITY:
Inclusion Criteria:

* Male and females 18-65 years old
* Generally healthy
* Able to provide informed consent
* Recent positive COVID-19 test (per RT-PCR Test)*

Exclusion Criteria:

* Unstable or serious illness (e.g. kidney, liver, GIT, heart conditions, diabetes, thyroid gland function, malignancy, HIV, lung conditions or chronic asthma)
* Serious mood disorders, neurological disorders such as MS, or cognitive damage
* Active smokers and/or nicotine or drug abuse
* Active, regular marijuana or other cannabinoid use, other street/recreational drug use
* Chronic past and/or current alcohol use (>14 alcoholic drinks week)
* Allergic to any of the ingredients in active or placebo formula including peanuts, eggs or turmeric
* Pregnant or lactating woman
* People medically prescribed to take drugs that would affect the immune and/or the inflammatory response
* People who have had treatment (last 5 years) for cancer, or chronic use of steroids
* BMI >40

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
IL6 concentration | change from baseline at day 28
  interleukin-6

SECONDARY OUTCOMES:
serum CRP concentration | change from baseline at day 28
  C-reactive protein (high sensitivity)
serum ferritin concentration | change from baseline at day 28
  serum ferritin
serum ICAM concentration | change from baseline at day 28
  Intercellular Adhesion Molecule 1
serum NFk-beta concentration | change from baseline at day 28
  nuclear factor kappa-light-chain-enhancer of activated B cells
serum white blood cell differential | change from baseline at day 28
  white blood cell differential
serum p-selectin concentration | change from baseline at day 28
  cell adhesion molecule

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona Biomedical Collaborative, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fessler SN, Liu L, Chang Y, Yip T, Johnston CS. Palmitoylethanolamide Reduces Proinflammatory Markers in Unvaccinated Adults Recently Diagnosed with COVID-19: A Randomized Controlled Trial. J Nutr. 2022 Oct 6;152(10):2218-2226. doi: 10.1093/jn/nxac154. PMID 36084236